CLINICAL TRIAL: NCT03614247
Title: Cost-Effectiveness of Different Treatment Options for Lower Calyceal Stones of 1 to 2 Centimeters: A Prospective, Randomized Study
Brief Title: Cost-Effectiveness of Different Treatment Options for Lower Calyceal Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Training and Research Hospital (Other)
Collaborators: Ministry of Health, Turkey (Other Government)
Responsible Party: Principal Investigator, Muhammet Fatih Kilinc, Principal Investigator, Ankara Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2730
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-07

CONDITIONS: Renal Calculi
Keywords: Lower calyceal stone; cost-effectiveness; percutaneous nephrolithotomy; retrograde intrarenal surgery
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Intervention Model Description: Patients who had a lower calyceal stone between 1cm and 2cm in size
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- RIRS (Active Comparator): Patients underwent retrograde intrarenal surgery for lower calyceal stone between 1cm and 2cm in size
  Interventions: Procedure: Retrograde intrarenal surgery
- Micro-PNL (Active Comparator): Patients underwent micro percutaneous nephrolithotomy (tract size <10 F) for lower calyceal stone between 1cm and 2cm in size
  Interventions: Procedure: Micro-PNL
- Ultramini-PNL (Active Comparator): Patients underwent ultra-mini percutaneous nephrolithotomy (tract size <15 F) for lower calyceal stone between 1cm and 2cm in size
  Interventions: Procedure: Ultra-mini PNL
- Mini-PNL (Active Comparator): Patients underwent mini percutaneous nephrolithotomy (tract size <20 F) for lower calyceal stone between 1cm and 2cm in size
  Interventions: Procedure: Mini-PNL
- Standard PNL (Active Comparator): Patients underwent standard percutaneous nephrolithotomy (tract size >25 F) for lower calyceal stone between 1cm and 2cm in size
  Interventions: Procedure: Standard PNL

INTERVENTIONS:
Procedure: Retrograde intrarenal surgery — The procedure was performed with the patient in the dorsal lithotomy position under general anesthesia. Firstly, diagnostic ureteroscopy was done with a 6/7.5 Fr semi-rigid ureteroscope (Richard Wolf, Knittlingen, Germany). A 0.035mm double-tipped sensor guidewire was placed to the renal pelvis. A 10/12 Fr ureteric access sheath (Cook Medical, Indiana, USA) was used. A 7.5 Fr flexible ureteroscope (Flex X2, Karl Storz, Tuttlingen, Germany) was used for the main procedure. The stones were fragmented using a Holmium:Yttrium Aluminum Garnet laser (272 microns). At the end of each procedure, a double-j ureteric catheter and urethral catheter were routinely placed.
  Arms: RIRS
Procedure: Micro-PNL — The PNL procedures were performed with the patient in the prone position under general anesthesia. A 6-F ureteric catheter was placed at the beginning of the procedure. Calyceal access was provided using a 22-G Chiba needle. A 0.038mm sensor-tipped guidewire was inserted through the calyceal puncture into the renal pelvis. After tract dilatation, a sheath was inserted. The instruments used were a 4.8 Fr for micro PNL (PolyDiagnost, Pfaffenhofen, Germany). Stone fragmentation was carried out using laser in micro PNL. No nephrostomy was placed in any patient whom underwent micro PNL surgical technique. A double- j stent was placed in necessary (e.g., pelvis perforation, rest stone, stone migration to ureter). A urethral catheter was placed routinely in all patients.
  Arms: Micro-PNL
Procedure: Ultra-mini PNL — The PNL procedures were performed with the patient in the prone position under general anesthesia. A 6-F ureteric catheter was placed at the beginning of the procedure. Calyceal access was provided using a 22-G Chiba needle. A 0.038mm sensor-tipped guidewire was inserted through the calyceal puncture into the renal pelvis. After tract dilatation, a sheath was inserted. The instruments used were a 7.5 Fr for ultramini PNL (Karl Storz, Tuttlingen, Germany). Stone fragmentation was carried out using laser in ultramini PNL. No nephrostomy was placed in any patient whom underwent ultramini PNL surgical technique. A double- j stent was placed in necessary (e.g., pelvis perforation, rest stone, stone migration to ureter). A urethral catheter was placed routinely in all patients.
  Arms: Ultramini-PNL
Procedure: Mini-PNL — The PNL procedures were performed with the patient in the prone position under general anesthesia. A 6-F ureteric catheter was placed at the beginning of the procedure. Calyceal access was provided using a 22-G Chiba needle. A 0.038mm sensor-tipped guidewire was inserted through the calyceal puncture into the renal pelvis. After tract dilatation, a sheath was inserted. The instruments used were a 12 Fr for mini PNL (Karl Storz, Tuttlingen, Germany). Stone fragmentation was carried out using pneumatic, ultrasonic or laser in mini PNL. No nephrostomy was placed in any patient whom underwent mini PNL surgical technique. A double- j stent was placed in necessary (e.g., pelvis perforation, rest stone, stone migration to ureter). A urethral catheter was placed routinely in all patients.
  Arms: Mini-PNL
Procedure: Standard PNL — The PNL procedures were performed with the patient in the prone position under general anesthesia. A 6-F ureteric catheter was placed at the beginning of the procedure. Calyceal access was provided using a 22-G Chiba needle. A 0.038mm sensor-tipped guidewire was inserted through the calyceal puncture into the renal pelvis. After tract dilatation, a sheath was inserted. The instruments used were a 24 Fr for standard PNL (Karl Storz, Tuttlingen, Germany). Stone fragmentation was carried out using pneumatic, ultrasonic or laser in standard PNL. A nephrostomy was placed in all standard PNL patients at the end of the procedure
  Arms: Standard PNL

SUMMARY:
The aim of the present study to perform a full cost analysis for the complete clearance of calyceal stones by retrograde intrarenal surgery (RIRS) and percutaneous nephrolithotomy (PNL) for the treatment of lower calyceal stones between 1 and 2 centimeters (cm) in size.

DETAILED DESCRIPTION:
The lifelong prevalence of urinary system stone disease is approximately 15%. The lower calyx is the most common location where renal calculi occur. Because anatomical factors preclude spontaneous passage in this area, the need for treatment is more likely in lower calyceal stones. The European Association of Urology (EAU) suggests percutaneous nephrolithotomy (PNL) for stones larger than 2 centimeters (cm) and shock wave lithotripsy (SWL) or retrograde intrarenal surgery (RIRS) for stones smaller than 1cm as a first option, but controversy continues regarding the best treatment option for medium-sized lower calyceal stones of between 1cm and 2cm.

Medical costs are divided into two components: direct and indirect. Direct costs encompass all medical expenditures (e.g., drugs, hospital bed, all consumable and non-consumable materials used during the operation), while indirect costs include loss of working days for the patient. The stone-free rates (SFR) are reported as approximately 60% and 90% for one session of RIRS and PNL, respectively; however, no physician can guarantee a 100% SFR for one session. For this reason, a full cost analysis must include the direct and indirect costs of both the first and all auxiliary procedures.

The aim of this study was to perform a full cost analysis for the complete clearance of calyceal stones by RIRS and all PNL types for the treatment of lower calyceal stones between 1cm and 2cm in size.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had a lower calyceal stone between 1cm and 2 cm in size

Exclusion Criteria:

* solitary or anomaly (horseshoe or pelvic kidney) kidney,
* renal insufficiency,
* pregnancy,
* patient younger than 18 or older than 75 years,
* non-interrupted antithrombotic medication before surgery,
* urinary tract infection,
* double-j or nephrostomy insertion before surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Stone free status | 3 months
  Stone-free was defined as no rest stone or ≤ 3mm clinical insignificance rest stone

CONTACTS AND LOCATIONS:
Overall Officials: Muhammet F Kilinc, M.D., Principal Investigator — Ankara Training and Research Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Schoenthaler M, Wilhelm K, Hein S, Adams F, Schlager D, Wetterauer U, Hawizy A, Bourdoumis A, Desai J, Miernik A. Ultra-mini PCNL versus flexible ureteroscopy: a matched analysis of treatment costs (endoscopes and disposables) in patients with renal stones 10-20 mm. World J Urol. 2015 Oct;33(10):1601-5. doi: 10.1007/s00345-015-1489-4. Epub 2015 Jan 23. PMID 25614255
- [Result] Sabnis RB, Ganesamoni R, Doshi A, Ganpule AP, Jagtap J, Desai MR. Micropercutaneous nephrolithotomy (microperc) vs retrograde intrarenal surgery for the management of small renal calculi: a randomized controlled trial. BJU Int. 2013 Aug;112(3):355-61. doi: 10.1111/bju.12164. PMID 23826843
- [Result] Demirbas A, Resorlu B, Sunay MM, Karakan T, Karagoz MA, Doluoglu OG. Which Should be Preferred for Moderate-Size Kidney Stones? Ultramini Percutaneous Nephrolithotomy or Retrograde Intrarenal Surgery? J Endourol. 2016 Dec;30(12):1285-1289. doi: 10.1089/end.2016.0370. PMID 27706948